CLINICAL TRIAL: NCT05992662
Title: Mindfulness-Based Training Program in Bariatric Surgery Patients: An Action Research
Brief Title: Minfulness-Based Training Program in Bariatric Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Defne Dizlek, Research Asssistant, Akdeniz University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AkdenizBariatricSurgery
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Bariatric Surgery Candidate
Keywords: bariatric surgery; mindfulness; mindful eating; training program; surgery nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In this research, the training program was designed as an intervention.
  Summary of the research's implementation plan:
  Preparation of Mindfulness-based training program in bariatric surgery Inviting adult individuals to participate in the research before bariatric surgery and reaching the targeted number of participants Participants who agreed to participate in the study fill out the individual introduction form, complete the short story, and administer the Mindful Eating Questionnaire to the participants Conducting mindfulness-based 4-session training program Focus group discussion after the training Reminder of weekly practices Recording changes in mindful eating in participant experience diaries during the follow-up At the end of the monitoring phase (3rd-6th months), individual in-depth interviews and Mindful Eating Questionnaires are conducted with each participant in the action group
  Interventions: Behavioral: Mindfulness-Based Training Programme in Bariatric Surgey Patients
- Control Group (No Intervention): Mindful Eating Questionnaire will be applied before the surgery, at the 3rd and 6th months after the surgery. No intervention will be applied to the control group.

INTERVENTIONS:
Behavioral: Mindfulness-Based Training Programme in Bariatric Surgey Patients — ACTION Conducting mindfulness-based 4-session training program Focus group discussion after the training Within the scope of mindfulness-based training: Mindful Eating practices; qigong exercises; meditation exercises; breathing exercises; training specific to the bariatric surgery process was given.
  FOLLOW-UP PHASE (3rd MONTH/6.MONTH POSTOPERATIVE)
  * Reminder of weekly practices
  * Recording changes in mindful eating in participant experience diaries during the follow-up
  Arms: Intervention Group

SUMMARY:
Bariatric surgery maintains its place in the literature as the most effective treatment method for obesity. In order for the surgery to be effective, it is important for individuals to adapt to the surgical process. This process has become more manageable with lifestyle changes and health education. Mindfulness practices are (useful forms of intervention) for practicing and restructuring the brain for healthier eating habits. The results of mindfulness studies show that mindful eating practices can be effective in the prevention and treatment of obesity. Studies on mindfulness in obesity are increasing rapidly in the literature; however, few studies have tested this approach in bariatric surgery patients. This research was planned in an action research design to examine the effect of mindfulness-based education program on individuals' mindful eating in bariatric surgery patients. As an action in the research, an mindfullness-based training program will be developed for the bariatric patient group. Then, in the preoperative period, a four-week, weekly session of mindfulness-based exercise and eating training will be given to the action group as an intervention. Mindful Eating Questionnaire will be applied to all participants (action and control group) before the training, and data will be collected from the action group with the vignette technique. A short cut story will be prepared, and the participants will be asked to complete the short story in written form. At the end of the training sessions, a focus group discussion will be held with the participants. An in-depth interview will be conducted with each participant in line with the semi-structured interview form in the third and sixth months after the surgery. The Mindful Eating Questionnaire will be readministered to both the action group and the control group. During and after the training, participants will be asked to write down any changes they notice in their diaries. In the research, quantitative data will be evaluated with descriptive statistical tests, and qualitative data will be evaluated with content analysis, descriptive and thematic analysis. As a result of the research, it is aimed to improve the mindful eating of the participants. It is anticipated that the research will increase the mindfulness level of the participants in their lives and contribute to future research.

DETAILED DESCRIPTION:
This research was planned in an action research design to examine the effect of mindfulness-based training program on individuals' mindful eating in bariatric surgery patients. As an action in the research, an mindfullness-based training program will be developed for the bariatric patient group. Then, in the preoperative period, a four-week, weekly session of mindfulness-based exercise and eating training will be given to the action group as an intervention. Mindful Eating Questionnaire will be applied to all participants (action and control group) before the training, and data will be collected from the action group with the vignette technique. A short cut story will be prepared, and the participants will be asked to complete the short story in written form. At the end of the training sessions, a focus group discussion will be held with the participants. An in-depth interview will be conducted with each participant in line with the semi-structured interview form in the third and sixth months after the surgery. The Mindful Eating Questionnaire will be readministered to both the action group and the control group. During and after the training, participants will be asked to write down any changes they notice in their diaries. In the research, quantitative data will be evaluated with descriptive statistical tests, and qualitative data will be evaluated with content analysis, descriptive and thematic analysis. As a result of the research, it is aimed to improve the mindful eating of the participants. It is anticipated that the research will increase the mindfulness level of the participants in their lives and contribute to future research.

In this research, the training program was designed as an intervention. The training program consists of preparation, implementation, follow-up, and evaluation phases. The implementation plan of the research is summarized below:

PREPARATION PHASE Preparation of Mindfulness-based training program in bariatric surgery Inviting adult individuals to participate in research before bariatric surgery and reaching the targeted number of participants.

* Participants who agreed to participate in the study should fill out the individual introduction form, complete the cut short story, and apply the Mindful Eating Questionnaire to the participants.
* Application of the Mindful Eating Questionnaire to the Control Group

ACTION

* Conducting mindfulness-based 4-session training program
* Focus group discussion after the training

FOLLOW-UP PHASE (3rd MONTH/6.MONTH POSTOPERATIVE)

* Reminder of weekly practices
* Recording changes in mindful eating in participant experience diaries during the follow-up

DATA COLLECTION

* Individual in-depth interviews with each of the participants in the action group at the end of the follow-up phase (3rd and 6th months)
* At the end of the follow-up period, re-administration of the Mindful Eating Questionnaire to both the action and control groups (3rd and 6th months)

ELIGIBILITY:
Inclusion Criteria:

* People who agreed to participate in the research.
* Being included in the bariatric surgery list
* Over 18 years of age old
* Able to understand, speak and write Turkish.
* No cognitive problem in self-expression
* To be able to use the WhatsApp application effectively.
* Absence of alcohol or substance abuse
* No diagnosed psychotic and depressive disorder

Exclusion Criteria:

* Declaring that he will not continue the research at any stage of the research
* Not participating in the entire training program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Mindful Eating | Before the surgery, 3. and 6. Months after the surgery
  Mindful Eating Questionnaire There are 5 sub-factors in a 4-point Likert-type scale with 28 questions, the original name of which is the Mindful Eating Questionnaire (MEQ). The association between MEQ and eating behavior and emotional state can be carefully questioned. MEQ has been proposed by Framson et al. (2009) as a useful weight loss tool that has created non-judgmental awareness of physical and emotional sensations associated with eating. The validity and reliability analyze of the Mindful Eating Questionnaire (MEQ) for the Turkish sample were performed by Köse et al.

CONTACTS AND LOCATIONS:
Overall Officials: Defne Dizlek Bayraktar, Principal Investigator — Akdeniz University; Emine Catal, Study Chair — Akdeniz University; Huseyin Ciyiltepe, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Konyaalti, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abiles V, Rodriguez-Ruiz S, Abiles J, Mellado C, Garcia A, Perez de la Cruz A, Fernandez-Santaella MC. Psychological characteristics of morbidly obese candidates for bariatric surgery. Obes Surg. 2010 Feb;20(2):161-7. doi: 10.1007/s11695-008-9726-1. Epub 2008 Oct 29. PMID 18958537
- [Background] Baig SJ, Priya P, Mahawar KK, Shah S; Indian Bariatric Surgery Outcome Reporting (IBSOR) Group. Weight Regain After Bariatric Surgery-A Multicentre Study of 9617 Patients from Indian Bariatric Surgery Outcome Reporting Group. Obes Surg. 2019 May;29(5):1583-1592. doi: 10.1007/s11695-019-03734-6. PMID 30729366
- [Background] Caldwell AE, Purcell SA, Gray B, Smieja H, Catenacci VA. The impact of yoga on components of energy balance in adults with overweight or obesity: A systematic review. Obes Sci Pract. 2021 Aug 19;8(2):219-232. doi: 10.1002/osp4.552. eCollection 2022 Apr. PMID 35388342
- [Background] Carbone F, Adami G, Liberale L, Bonaventura A, Bertolotto M, Andraghetti G, Scopinaro N, Camerini GB, Papadia FS, Cordera R, Dallegri F, Montecucco F. Serum levels of osteopontin predict diabetes remission after bariatric surgery. Diabetes Metab. 2019 Sep;45(4):356-362. doi: 10.1016/j.diabet.2018.09.007. Epub 2018 Sep 27. PMID 30268840
- [Background] Chacko SA, Yeh GY, Davis RB, Wee CC. A mindfulness-based intervention to control weight after bariatric surgery: Preliminary results from a randomized controlled pilot trial. Complement Ther Med. 2016 Oct;28:13-21. doi: 10.1016/j.ctim.2016.07.001. Epub 2016 Jul 12. PMID 27670865
- [Background] Dunn C, Haubenreiser M, Johnson M, Nordby K, Aggarwal S, Myer S, Thomas C. Mindfulness Approaches and Weight Loss, Weight Maintenance, and Weight Regain. Curr Obes Rep. 2018 Mar;7(1):37-49. doi: 10.1007/s13679-018-0299-6. PMID 29446036
- [Background] Lauti M, Kularatna M, Hill AG, MacCormick AD. Weight Regain Following Sleeve Gastrectomy-a Systematic Review. Obes Surg. 2016 Jun;26(6):1326-34. doi: 10.1007/s11695-016-2152-x. PMID 27048439
- [Background] Leung KW, Yang YJ, Hui SS, Woo J. Mind-Body Health Benefits of Traditional Chinese Qigong on Women: A Systematic Review of Randomized Controlled Trials. Evid Based Complement Alternat Med. 2021 Sep 14;2021:7443498. doi: 10.1155/2021/7443498. eCollection 2021. PMID 34567220
- [Background] Liu T, Bai S, Zhang RC. [Effects of Health Qigong Baduanjin on diabetes related indexes in middle-aged obese women]. Zhongguo Ying Yong Sheng Li Xue Za Zhi. 2018 Jan 8;34(1):19-22. doi: 10.12047/j.cjap.5484.2018.006. Chinese. PMID 29926653
- [Background] Lyzwinski LN, Caffery L, Bambling M, Edirippulige S. The Mindfulness App Trial for Weight, Weight-Related Behaviors, and Stress in University Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Apr 10;7(4):e12210. doi: 10.2196/12210. PMID 30969174
- [Background] Mason AE, Jhaveri K, Cohn M, Brewer JA. Testing a mobile mindful eating intervention targeting craving-related eating: feasibility and proof of concept. J Behav Med. 2018 Apr;41(2):160-173. doi: 10.1007/s10865-017-9884-5. Epub 2017 Sep 16. PMID 28918456
- [Background] Miller-Matero LR, Bryce K, Saulino CK, Dykhuis KE, Genaw J, Carlin AM. Problematic Eating Behaviors Predict Outcomes After Bariatric Surgery. Obes Surg. 2018 Jul;28(7):1910-1915. doi: 10.1007/s11695-018-3124-0. PMID 29417489
- [Background] Palacio A, Luna C, Maiz C, Blanco E. Nutritional and behavioral factors related to weight gain after bariatric surgery. Rev Med Chil. 2021 Jan;149(1):30-36. doi: 10.4067/S0034-98872021000100030. PMID 34106133
- [Background] Sairanen E, Tolvanen A, Karhunen L, Kolehmainen M, Jarvela E, Rantala S, Peuhkuri K, Korpela R, Lappalainen R. Psychological flexibility and mindfulness explain intuitive eating in overweight adults. Behav Modif. 2015 Jul;39(4):557-79. doi: 10.1177/0145445515576402. Epub 2015 Mar 25. PMID 25810381
- [Background] Sarwer DB, Dilks RJ, West-Smith L. Dietary intake and eating behavior after bariatric surgery: threats to weight loss maintenance and strategies for success. Surg Obes Relat Dis. 2011 Sep-Oct;7(5):644-51. doi: 10.1016/j.soard.2011.06.016. Epub 2011 Jul 13. PMID 21962227
- [Background] Siu PM, Yu AP, Chin EC, Yu DS, Hui SS, Woo J, Fong DY, Wei GX, Irwin MR. Effects of Tai Chi or Conventional Exercise on Central Obesity in Middle-Aged and Older Adults : A Three-Group Randomized Controlled Trial. Ann Intern Med. 2021 Aug;174(8):1050-1057. doi: 10.7326/M20-7014. Epub 2021 Jun 1. PMID 34058100
- [Background] Warren JM, Smith N, Ashwell M. A structured literature review on the role of mindfulness, mindful eating and intuitive eating in changing eating behaviours: effectiveness and associated potential mechanisms. Nutr Res Rev. 2017 Dec;30(2):272-283. doi: 10.1017/S0954422417000154. Epub 2017 Jul 18. PMID 28718396
- [Background] Zunker C, Karr T, Saunders R, Mitchell JE. Eating behaviors post-bariatric surgery: a qualitative study of grazing. Obes Surg. 2012 Aug;22(8):1225-31. doi: 10.1007/s11695-012-0647-7. PMID 22527594
- [Background] Tsai C, Steffen R, Kessler U, Merki H, Zehetner J. Short-term outcomes of endoscopic gastro-jejunal revisions for treatment of dumping syndrome after Roux-En-Y gastric bypass. Surg Endosc. 2020 Aug;34(8):3626-3632. doi: 10.1007/s00464-019-07137-7. Epub 2019 Sep 24. PMID 31552507
- [Background] Saunders R. "Grazing": a high-risk behavior. Obes Surg. 2004 Jan;14(1):98-102. doi: 10.1381/096089204772787374. PMID 14980042
- [Background] de Zwaan M, Hilbert A, Swan-Kremeier L, Simonich H, Lancaster K, Howell LM, Monson T, Crosby RD, Mitchell JE. Comprehensive interview assessment of eating behavior 18-35 months after gastric bypass surgery for morbid obesity. Surg Obes Relat Dis. 2010 Jan-Feb;6(1):79-85. doi: 10.1016/j.soard.2009.08.011. Epub 2009 Sep 3. PMID 19837012
- [Background] Czepczor-Bernat K, Brytek-Matera A, Gramaglia C, Zeppegno P. The moderating effects of mindful eating on the relationship between emotional functioning and eating styles in overweight and obese women. Eat Weight Disord. 2020 Aug;25(4):841-849. doi: 10.1007/s40519-019-00740-6. Epub 2019 Jul 16. PMID 31313253